CLINICAL TRIAL: NCT00351052
Title: A 24-Week, Randomized, Multicenter, Parallel-Group, Double-Blind, Vehicle-Controlled Study on Pimecrolimus Cream 1% Assessing the Steroid-Sparing Effect in the Long Term Management of Pediatric Patients With Severe Atopic Dermatitis
Brief Title: Steroid-Sparing Effect With Pimecrolimus in Pediatric Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981CDE10
Record Dates: First submitted 2006-07-10; First posted 2006-07-12 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Atopic Dermatitis
Keywords: Pimecrolimus, Atopic Dermatitis, Eczema, Pediatric
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Pimecrolimus
  Interventions: Drug: Pimecrolimus
- 2 (Placebo Comparator): Vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimecrolimus — Pimecroliums cream 1 % bid.
  Other Names: Elidel
  Arms: 1
Drug: Placebo — Vehicle control (placebo) bid.
  Arms: 2

SUMMARY:
This study will investigate the steroid sparing effect of pimecrolimus cream 1% in pediatric atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged 2 to < 18 years with severe AD (score 8 or 9 according to Rajka and Langeland)
* responded to 21 days of treatment with prednicarbate cream 0.25% during screening phase

Exclusion Criteria:

* Patients who had received phototherapy, systemic or topical therapy or systemic corticosteroids shortly prior to study

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 184 (Actual)
Dates: Start 2001-12; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Corticoid-sparing effect of pimecrolimus cream 1%

SECONDARY OUTCOMES:
atopic dermatitis control
safety of pimecrolimus cream 1%
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Novartis AG, Study Chair — Novartis
Locations (1):
- Investigational Site, Germany